CLINICAL TRIAL: NCT01878669
Title: Effects of N-acetyl Cysteine on Periprocedural Myocardial Infarction and Major Cardiac and Cerebral Events in Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Effects of N-acetyl Cysteine During Percutaneous Coronary Intervention
Acronym: EASE-PCI
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mehmet Ozaydin, MD, MD, Professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ozaydin289
Record Dates: First submitted 2013-03-26; First posted 2013-06-17 (Estimated); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: n-acetyl cysteine; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Acetylcysteine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- saline (Placebo Comparator): 30 mg/kg/15 min intravenous bolus preprocedural and 50 mg/kg/8 h intravenous infusion during and after the procedure
  Interventions: Drug: Saline
- n-acetyl cysteine (Experimental): 30 mg/kg/15 min intravenous bolus preprocedural and 50 mg/kg/8 h intravenous infusion during and after the procedure
  Interventions: Drug: N-acetyl cysteine

INTERVENTIONS:
Drug: N-acetyl cysteine
  Arms: n-acetyl cysteine
Drug: Saline
  Arms: saline

SUMMARY:
The aim of this study is to evaluate the effects of N-acetyl cysteine on periprocedural myocardial infarction and major cardiac and cerebral events in patients undergoing percutaneous coronary intervention and who have moderate to high risk for contrast induced nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old undergoing percutaneous coronary intervention and who have moderate to high risk for contrast induced nephropathy (Mehran Score ≥ 5)

Exclusion Criteria:

* Primary percutaneous coronary intervention
* Low risk for contrast induced nephropathy (Mehran Score < 5)
* Use of nephrotoxic agents (NSAIDs, aminoglycosides,recent contrast injection...)
* Infection
* Pregnancy, Lactation
* Renal failure requiring dialysis
* Hepatic failure
* History allergy for NAC
* History of Asthma
* Chronic nitrate usage
* Malignancy
* Use of corticosteroids
* Leukocytosis,Thrombocytosis,Anemia
* Blood pressure of >180/100mmHg despite anti-hypertensive therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-09 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
periprocedural myocardial infarction | postprocedural 3-6 h

SECONDARY OUTCOMES:
NAC side effects (Asthma exacerbation, pruritus, dyspnea) | during hospitalization at 48 hours
major cardiac and cerebral events | 1 year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University, Isparta, Mediterranean Region, Turkey (Türkiye)